CLINICAL TRIAL: NCT05537870
Title: The Effectiveness of Nurse Navigators in Cancer Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Chang, Hsiu-Ju, professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201809031
Record Dates: First submitted 2022-08-29; First posted 2022-09-13 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Neoplasms; Nurse-Patient Relations; Psychiatric Disorder
Keywords: Navigator
MeSH Terms: conditions — Neoplasms; Mental Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Eligible patient were randomly assigned by the computer random number generator to either intervention or control group. Several methods were used to maintain the treatment blindly, including segregation of assessment and treatment staff and instructions to patients to avoid discussion of treatment assignment with the independent evaluators.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cancer navigator care (Active Comparator): experimental group: case manager care combined cancer nurse navigator care
  Interventions: Behavioral: cancer nurse navigator care
- case manager care (Placebo Comparator): control group: only case manager care(usual care)
  Interventions: Behavioral: case manager care

INTERVENTIONS:
Behavioral: cancer nurse navigator care — oncology case manager care combined with cancer nurse navigator care
  Arms: cancer navigator care
Behavioral: case manager care — case manager care (usual care)
  Arms: case manager care

SUMMARY:
Cancer patients will be recruited from the Taipei Cancer Center of Taipei Medical University. This study was divided into two phases. The first phase adopted cross-sectional study design with questionnaires to analyze the potential predictors of depressive symptoms among cancer patients. The second stage was adopted experimental study design to explore the effectiveness of nurse navigators in cancer care.

DETAILED DESCRIPTION:
The first phase analyze the potential predictors include the following: socio-demographic characteristics, disease characteristics, lifestyle, perceived benefits, cancer patient' experience with medical service, emotional distress, anxiety, and demoralization.

The second phase will be experimental study.Thus, subjects were randomly sampled and divided into 2 groups: experimental group and control group. Subjects in the experimental group will receive oncology case manager care combined with cancer nurse navigator care, while subjects in the control group will be designed as regular care, which only care with cancer case managers. Both groups will receive long-term follow-up analysis (pre-intervention, post-intervention - 3 months, and 6 months). Outcome measures include the following: perceived benefits, emotional distress, depression and anxiety, demoralization, cancer patient' experience with medical service, and medical report indicators (retention rate, completion rate, survival rate, mortality rate, untreated cancer within 3 months).

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients for the first time at the cancer center clinic of the university hospital
2. Older than 20 years old
3. Ability to communicate and read
4. The case voluntarily participated in the study and signed the consent form

Exclusion Criteria:

1. People with mental disorders who have schizophrenia, personality disorder, mental retardation, or organic brain disorder.
2. Patient with brain metastasis.
3. Patients who receive hospice palliative care or other treatment programs.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Perceived benefits scale (PBS), questionnaires to measure self-efficacy | Mainly consists of repeated measurements at three time points (Baseline, 3th month, and 6th month). Changes in scores on the PBS questionnaire after intervention were assessed using baseline scores as reference values.
  Questionnaires to measure self-efficacy collected at three time points (baseline, 3th month, and 6th month). Evaluate the effectiveness of interventions in PBS at three time points.
The Patient Assessment of Chronic Illness Care (PACIC), questionnaires to measure patient' experience | Mainly consists of repeated measurements at three time points (Baseline, 3th month, and 6th month). Changes in scores on the PACIC questionnaire after intervention were assessed using baseline scores as reference values.
  Questionnaires to measure patient' experience with medical service collected at three time points (baseline, 3th month, and 6th month). Evaluate the effectiveness of interventions in PACIC at three time points.
Distress Thermometer and Problem List (DT), questionnaires to measure emotional distress and psychological problems | Mainly consists of repeated measurements at three time points (baseline, 3th month, and 6th month). Changes in scores on the DT questionnaire after intervention were assessed using baseline scores as reference values.
  Questionnaires to measure emotional distress and psychological problems collected at three time points (baseline, 3th month, and 6th month). Evaluate the effectiveness of interventions in DT at three time points.
Hospital Anxiety and Depression Scale (HADS), questionnaires to measure anxiety and depression | Mainly consists of repeated measurements at three time points (baseline, 3th month, and 6th month). Changes in scores on the HADS questionnaire after intervention were assessed using baseline scores as reference values.
  Questionnaires to measure anxiety and depression collected at three time points (baseline, 3th month, and 6th month). Evaluate the effectiveness of interventions in HADS at three time points.
Demoralization Scale- Mandarin Version (DS-MV), questionnaires to measure demoralization | Mainly consists of repeated measurements at three time points (baseline, 3th month, and 6th month). Changes in scores on the DS-MV questionnaire after intervention were assessed using baseline scores as reference values.
  Questionnaires to measure demoralization collected at three time points (baseline, 3th month, and 6th month). Evaluate the effectiveness of interventions in HADS at three time points.

SECONDARY OUTCOMES:
The retention rate | At the sixth month, statistical analysis was performed based on the report indicators of the retention rate obtained from the hospital medical record information.
  Medical report indicators of the retention rate collected at 6th month
The completion rate | At the sixth month, statistical analysis was performed based on the report indicators of the completion rate obtained from the hospital medical record information.
  Medical report indicators of the completion rate collected at 6th month
The survival rate | At the sixth month, statistical analysis was performed based on the report indicators of the survival rate obtained from the hospital medical record information.
  Medical report indicators of the survival rate collected at 6th month
The mortality rate | At the sixth month, statistical analysis was performed based on the report indicators of the mortality rate obtained from the hospital medical record information.
  Medical report indicators of the mortality rate collected at 6th month
The untreated rate of cancer within 3 months | At the sixth month, statistical analysis was performed based on the report data of the untreated rate of cancer within 3 months obtained from the hospital medical record information
  Medical report indicators of the untreated rate of cancer within 3 months collected at 6th month

CONTACTS AND LOCATIONS:
Overall Officials: hsiu-ju Chang, PhD, Study Chair — Taipei Medical Unviersity
Locations (1):
- Wan Fang Hospital, Taipei Medical University, Taipei, Wenshan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitchell AJ, Chan M, Bhatti H, Halton M, Grassi L, Johansen C, Meader N. Prevalence of depression, anxiety, and adjustment disorder in oncological, haematological, and palliative-care settings: a meta-analysis of 94 interview-based studies. Lancet Oncol. 2011 Feb;12(2):160-74. doi: 10.1016/S1470-2045(11)70002-X. Epub 2011 Jan 19. PMID 21251875
- [Result] Allemani C, Matsuda T, Di Carlo V, Harewood R, Matz M, Niksic M, Bonaventure A, Valkov M, Johnson CJ, Esteve J, Ogunbiyi OJ, Azevedo E Silva G, Chen WQ, Eser S, Engholm G, Stiller CA, Monnereau A, Woods RR, Visser O, Lim GH, Aitken J, Weir HK, Coleman MP; CONCORD Working Group. Global surveillance of trends in cancer survival 2000-14 (CONCORD-3): analysis of individual records for 37 513 025 patients diagnosed with one of 18 cancers from 322 population-based registries in 71 countries. Lancet. 2018 Mar 17;391(10125):1023-1075. doi: 10.1016/S0140-6736(17)33326-3. Epub 2018 Jan 31. PMID 29395269
- [Result] Burgess C, Cornelius V, Love S, Graham J, Richards M, Ramirez A. Depression and anxiety in women with early breast cancer: five year observational cohort study. BMJ. 2005 Mar 26;330(7493):702. doi: 10.1136/bmj.38343.670868.D3. Epub 2005 Feb 4. PMID 15695497
- [Result] Glasgow RE, Wagner EH, Schaefer J, Mahoney LD, Reid RJ, Greene SM. Development and validation of the Patient Assessment of Chronic Illness Care (PACIC). Med Care. 2005 May;43(5):436-44. doi: 10.1097/01.mlr.0000160375.47920.8c. PMID 15838407
- [Result] Hoffman BM, Zevon MA, D'Arrigo MC, Cecchini TB. Screening for distress in cancer patients: the NCCN rapid-screening measure. Psychooncology. 2004 Nov;13(11):792-9. doi: 10.1002/pon.796. PMID 15386639
- [Result] Kissane DW, Wein S, Love A, Lee XQ, Kee PL, Clarke DM. The Demoralization Scale: a report of its development and preliminary validation. J Palliat Care. 2004 Winter;20(4):269-76. PMID 15690829
- [Result] Lee CY, Fang CK, Yang YC, Liu CL, Leu YS, Wang TE, Chang YF, Hsieh RK, Chen YJ, Tsai LY, Liu SI, Chen HW. Demoralization syndrome among cancer outpatients in Taiwan. Support Care Cancer. 2012 Oct;20(10):2259-67. doi: 10.1007/s00520-011-1332-4. Epub 2011 Nov 27. PMID 22120003
- [Result] Linden W, Vodermaier A, Mackenzie R, Greig D. Anxiety and depression after cancer diagnosis: prevalence rates by cancer type, gender, and age. J Affect Disord. 2012 Dec 10;141(2-3):343-51. doi: 10.1016/j.jad.2012.03.025. Epub 2012 Jun 21. PMID 22727334
- [Result] Lynch MP, Cope DG, Murphy-Ende K. Advanced practice issues: results of the ONS Advanced Practice Nursing survey. Oncol Nurs Forum. 2001 Nov-Dec;28(10):1521-30. PMID 11759300
- [Result] Moorey S, Greer S, Watson M, Gorman C, Rowden L, Tunmore R, Robertson B, Bliss J. The factor structure and factor stability of the hospital anxiety and depression scale in patients with cancer. Br J Psychiatry. 1991 Feb;158:255-9. doi: 10.1192/bjp.158.2.255. PMID 1812841
- [Result] Neilson KA, Pollard AC, Boonzaier AM, Corry J, Castle DJ, Mead KR, Gray MC, Smith DI, Trauer T, Couper JW. Psychological distress (depression and anxiety) in people with head and neck cancers. Med J Aust. 2010 Sep 6;193(S5):S48-51. doi: 10.5694/j.1326-5377.2010.tb03928.x. PMID 21542446
- [Result] Roth AJ, Kornblith AB, Batel-Copel L, Peabody E, Scher HI, Holland JC. Rapid screening for psychologic distress in men with prostate carcinoma: a pilot study. Cancer. 1998 May 15;82(10):1904-8. doi: 10.1002/(sici)1097-0142(19980515)82:103.0.co;2-x. PMID 9587123
- [Result] Wang GL, Hsu SH, Feng AC, Chiu CY, Shen JF, Lin YJ, Cheng CC. The HADS and the DT for screening psychosocial distress of cancer patients in Taiwan. Psychooncology. 2011 Jun;20(6):639-46. doi: 10.1002/pon.1952. Epub 2011 Mar 15. PMID 21626611
- [Result] O'Connor M, White K, Kristjanson LJ, Cousins K, Wilkes L. The prevalence of anxiety and depression in palliative care patients with cancer in Western Australia and New South Wales. Med J Aust. 2010 Sep 6;193(S5):S44-7. doi: 10.5694/j.1326-5377.2010.tb03927.x. PMID 21542445
- [Result] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- See also: cancer — http://www.who.int/mediacentre/factsheets/fs297/en/.